CLINICAL TRIAL: NCT06571500
Title: Growth Hormone Resistance of Beta-cells in People With a Family History of Type 2 Diabetes
Brief Title: Growth Hormone Resistance of Beta-cells in Women and People
Acronym: GHRB-B
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research; Professor, Medicine & Nutrition; NextGen Director of Clinical and Translational Sciences Unit, University of Missouri-Columbia
Other Study IDs: 2111127-B
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Men and women with a family history of type 2 diabetes
- Men and women without a family history of type 2 diabetes

SUMMARY:
The purpose of the research study is to better understand how beta-cells (cells in the pancreas that make insulin and help regulate blood sugar) respond to growth hormone in people with a family history of type 2 diabetes at the University of Missouri. Our aim is to advance understanding of how growth hormone affects beta-cells and risk factors for developing gestational diabetes and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* hemoglobin HbA1c ≤5.6% and fasting blood glucose <100 mg/dl
* body mass index ≥30.0 kg/m2 and <45.0 kg/m2

Additional, group-specific inclusion criteria:

* Family history of type 2 diabetes: first degree relative with type 2 diabetes
* Control group: no family history of type 2 diabetes

Exclusion Criteria:

* Pregnant, planning to become pregnant during the study, or breastfeeding
* Current diagnosis or history of type 1 or type 2 diabetes
* Use of medications that can impact the study outcomes (e.g., GLP-1 receptor agonists)
* History of bariatric surgery
* Known hypothyroidism or use of thyroid medications
* History of intracranial hypertension, including papilledema, or a condition that increases the risk of developing intracranial hypertension, such as Turner Syndrome, Prader-Willi Syndrome, or renal impairment
* Current cancer or cancer that has been in remission less than 5 years
* First degree relative with type 1 diabetes diagnosis
* Evidence of significant anemia or significant end organ dysfunction (e.g., liver, kidney, heart disease)
* Alcohol use disorder, use of controlled substances, or smoking >2 cigarettes per day
* Greater than 3% weight loss within three months of screening or engaged in regular (≥3 days per week), continuous moderate- or high-intensity exercise of ≥30 min duration
* Mentally disabled persons, prisoners, and persons with inability to grant voluntary informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of obese men and women ages 18-45 with and without a first degree relative with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Beta-cell function | 15, 30, 60, 120, 240, and 360 min and 7 days after rhGH administration
  Insulin secretion rate in relationship to plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No